CLINICAL TRIAL: NCT03601468
Title: Association Between Autism and Iron Deficiency in Children Diagnosed Autism
Brief Title: Association Between Autism and Iron Deficiency
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Ali Mohammed Mostafa, Assiut university, Assiut University
Other Study IDs: Assiut university 2018
Record Dates: First submitted 2018-07-08; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Autism in Children
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Association between Autism and Iron Deficiency in Children Diagnosed Autism

DETAILED DESCRIPTION:
Autism is a behaviorally defined complex neurodevelopmental syndrome characterized by impairments in social communication, by the presence of restricted and repetitive behaviors, interests and activities, and by abnormalities in sensory reactivity.

Autism is a severe, life-long developmental disorder that compromises functioning across multiple domains including social behavior, language, sensory function, and ritualistic/repetitive behaviors and interests. While the etiology of autism is complex and not fully understood, strong evidence from twin and family studies suggests a large genetic contribution .

Autism is caused by a combination of genetic and environment factors. Risk factors include certain infections during pregnancy such as rubella as well as valproic acid, alcohol or cocaine use during pregnancy.

The number of children known to have autism has increased dramatically since the 1980's.The reviews of epidemiology in estimating the global prevalence is that one to two cases of autism exist per 2,000 people, and about six per 1,000 people have Autistic Spectrum Disorders (ASD) .

According to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), a guide created by the American Psychiatric Association used to diagnose mental disorders, people with Autism have:

* Difficulty with communication and interaction with other people
* Restricted interests and repetitive behaviors
* Symptoms that hurt the person's ability to function properly in school, work, and other areas of life.

Iron deficiency (ID) is the most common and persevering nutritional disorder and continues to be an important public health problem worldwide. Specifically in children in the first years of life, hemoglobin (HGB) levels below 11 g/dL have been related to negative cognitive, social, and emotional effects that may lead to irreversible behavioral squeals, even after appropriate treatment.

A reduction of iron levels in the brain may be accompanied by changes in serotonergic and dopaminergic systems, cortical networks, and myelination.

Iron deficiency (ID) cause negative outcomes on psychomotor and behavioral development of infants and young children. Children with autism are under risk for ID and this condition may increase the severity of psychomotor and behavioral problems,The association between iron deficiency and developmental problems such as global developmental delay is thought to be bidirectional. Iron deficiency impairs the processes of neurotransmitter metabolism and myelin formation, as well as altering energy metabolism in the brain - effects that have been theorised to cause behavioural and cognitive developmental delays in children.

Thus, it can be considered that ID/IDA (iron deficiency anemia) may increase the severity of autistic symptoms in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* All children with autism above 2 years to and do not take supplements of iron or vitamins.

Exclusion Criteria:

* • children less than 2 years old.

  * Children with other chronic neurological disorders or physical illness than Autism.
  * children with infection or other inflammatory conditions were excluded from the study,
  * children who received iron supplements during the last 3 months and / or who were on any dietary restrictions and children who are inpatients in rehabilitation centers

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Association between Autism and Iron Deficiency in Children Diagnosed Autism
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Aggressive autism picture | One year
  Identify the relationship between ID/IDA which may increase the severity of autistic symptoms in children with ASD.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Mohammed, Residant, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided